CLINICAL TRIAL: NCT06443944
Title: An Expanded Access Program of Cretostimogene Grenadenorepvec in Patients With Non-Muscle Invasive Bladder Cancer (NMIBC) Unresponsive to Bacillus Calmette-Guerin (BCG)
Brief Title: An Expanded Access Program of Cretostimogene Grenadenorepvec for Treatment of NMIBC for Patients Unresponsive to BCG
Status: Available | Type: Expanded Access
Sponsor: CG Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CRETO-EAP
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Non-Muscle Invasive Bladder Cancer; Urothelial Carcinoma; Urologic Cancer; Bladder Cancer
Keywords: Urology; Bladder Cancer; Non Muscle Invasive Bladder Cancer; Cretostimogene Grenadenorepvec
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Carcinoma, Transitional Cell; Urologic Neoplasms; Urinary Bladder Neoplasms | interventions — dodecyl maltoside

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Cretostimogene Grenadenorepvec — Engineered Oncolytic Adenovirus
  Other Names: CG0070
Other: n-dodecyl-B-D-maltoside — Transduction-enhancing agent
  Other Names: DDM

SUMMARY:
This is an open-label, expanded access trial designed to provide access to cretostimogene in patients with NMIBC (specifically CIS with or without HG Ta/T1) unresponsive to BCG.

DETAILED DESCRIPTION:
All participants will be assigned the same treatment schedule. Participants will receive an induction course of 6 weekly treatments, and, if there is no disease recurrence at Week 13, participants will receive a cycle of 3 weekly treatments up to Week 15.

If there is persistent HG Ta and/or CIS at Week 13, participants may receive a second induction cycle.

If the participant has persistent but improved HG Ta and/or CIS at Week 25 or a later timepoint, the participant may receive a cycle of 3 weekly treatments of cretostimogene at the discretion of the Investigator provided that T1 or higher stage of urothelial carcinoma is not present.

If there is no disease present at Week 25 or a later timepoint, participants will receive a cycle of 3 weekly treatments every 12 weeks through Month 12.

After Month 12, participants will receive a cycle of 3 weekly treatments every 6 months through the last treatment cycle at Month 24, or until discontinuation from the study treatment.

Disease status will be assessed based on local standard of care (which may include urine cytology, cystoscopy, and directed TURBT/biopsy) every 12 weeks. CTU/MRU can be done per standard of care evaluation at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Have pathologically confirmed BCG unresponsive CIS. There is no maximum limit to the amount of prior BCG treatment, but maintenance BCG should be administered on a schedule consistent with standard induction-maintenance protocols. Specifically, the definition of BCG unresponsive CIS will also require the following:

   * Pathologically confirmed relapsed or persistent CIS (with or without HG Ta or HG T1 disease)
   * Completion of qualifying BCG treatment (e.g., "5+2" minimum exposure) within 15 months of the initial qualifying dose of BCG.
2. Have all Ta and/or T1 disease and all CIS resected or fulgurated, as feasible, prior to study treatment
3. Ineligible to receive radical cystectomy (medically unfit) or refusal of radical cystectomy according to Investigator assessment.
4. Acceptable baseline organ function

Exclusion Criteria:

1. Muscle invasive bladder cancer, locally advanced or metastatic bladder cancer.
2. Has had active autoimmune or inflammatory disease requiring systemic treatment within 4 weeks of Day 1. Replacement therapy is not considered an excluded form of systemic treatment and is allowed.
3. Has received systemic anticancer therapy, including investigational agents, within 4 weeks of Day 1
4. Is pregnant, currently breastfeeding or intending to breastfeed, beginning at Screening through 1 week after the last study treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Michael G. Oefelein Clinical Trials, Bakersfield, California
  - McR, Llc., Murrieta, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Advanced Urology Institute, Daytona Beach, Florida
  - Advanced Urology Institute, Largo, Florida
  - Emory University, Atlanta, Georgia
  - Uropartners c/o Associated Urological Specialists, Chicago Ridge, Illinois
  - UroPartners, LLC, Glenview, Illinois
  - Urologic Specialists of Northwest Indiana, Merrillville, Indiana
  - Urology Center of Iowa Research, Clive, Iowa
  - Michigan Institute of Urology, PC, Troy, Michigan
  - The Urology Group, P.C., Southaven, Mississippi
  - Integrated Medical Professionals, PLLC, New York, New York
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Lowcountry Urology Clinics, PA, North Charleston, South Carolina
  - Urology Partners of North Texas Research Institute, Arlington, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology San Antonio, PA dba USA Clinical Trials, San Antonio, Texas
  - Digestive Health Research of North Texas, Wichita Falls, Texas
  - Spokane Urology, Spokane, Washington

REFERENCES:
- [Background] Chang SS, Boorjian SA, Chou R, Clark PE, Daneshmand S, Konety BR, Pruthi R, Quale DZ, Ritch CR, Seigne JD, Skinner EC, Smith ND, McKiernan JM. Diagnosis and Treatment of Non-Muscle Invasive Bladder Cancer: AUA/SUO Guideline. J Urol. 2016 Oct;196(4):1021-9. doi: 10.1016/j.juro.2016.06.049. Epub 2016 Jun 16. PMID 27317986
- [Background] Holzbeierlein JM, Bixler BR, Buckley DI, Chang SS, Holmes R, James AC, Kirkby E, McKiernan JM, Schuckman AK. Diagnosis and Treatment of Non-Muscle Invasive Bladder Cancer: AUA/SUO Guideline: 2024 Amendment. J Urol. 2024 Apr;211(4):533-538. doi: 10.1097/JU.0000000000003846. Epub 2024 Jan 24. PMID 38265030
- See also: NCCN Guidelines Bladder Cancer 1.2025 — https://www.nccn.org/guidelines/recently-published-guidelines